CLINICAL TRIAL: NCT02473510
Title: A Phase 4 Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety of 3 New 6:2 Influenza Virus Reassortants in Adults
Brief Title: Study to Evaluate the Safety of 3 New 6:2 Influenza Virus Reassortants in Adults for the 2015-2016 Season
Acronym: FluMist
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: D2560C00009
Record Dates: First submitted 2015-06-12; First posted 2015-06-16 (Estimated); Results first posted 2016-11-28 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-10

CONDITIONS: Influenza; Healthy
Keywords: Trivalent; Influenza; FluMist Quadrivalent; Vaccine; Prevention; Healthy
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Trivalent Influenza Vaccine (Experimental): A single dose of 10^(7.0 +/- 0.5) fluorescent focus units (FFU) per strain of trivalent influenza vaccine will be administered as intranasal spray on Day 1.
  Interventions: Biological: Trivalent Influenza Vaccine
- Placebo (Placebo Comparator): A single dose of placebo matched to trivalent influenza vaccine will be administered as intranasal spray on Day 1.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Trivalent Influenza Vaccine — A single dose of 10^(7.0 ± 0.5) FFU per strain of trivalent influenza vaccine will be administered as intranasal spray on Day 1.
  Arms: Trivalent Influenza Vaccine
Other: Placebo — A single dose of placebo matched to trivalent influenza vaccine will be administered as intranasal spray on Day 1.
  Arms: Placebo

SUMMARY:
This prospective annual release study is designed to evaluate the safety of 3 new influenza virus vaccine strains to be included in FluMist Quadrivalent for the 2015-2016 influenza season

DETAILED DESCRIPTION:
This prospective, randomized, double-blind, placebo-controlled release study will enroll approximately 300 healthy adults 18 to 49 years of age. Eligible participants will be randomly assigned in a 4:1 fashion to receive a single dose of trivalent vaccine or placebo by intranasal spray. Randomization will be stratified by site. This study will be conducted at 3 sites in the United States of America. Each participant will receive 1 dose of investigational product on Day 1. The duration of study participation for each participant is the time from study vaccination through 181 days after study vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 through 49 years
* Written informed consent
* Participant available by telephone
* Ability to understand and comply with the requirements of the protocol, as judged by the Investigator

Exclusion Criteria:

* Concurrent enrollment in another clinical study up to 180 days after receipt of investigational product (Day 181)
* History of hypersensitivity to any component of the vaccine, including egg or egg protein or serious, life threatening, or severe reactions to previous influenza vaccinations
* Any condition for which the inactivated influenza vaccine is indicated, including chronic disorders of the pulmonary or cardiovascular systems (example [eg], asthma), chronic metabolic diseases (eg, diabetes mellitus), renal dysfunction, or hemoglobinopathies that required regular medical follow-up or hospitalization during the preceding year
* Acute febrile (greater than [>] 100.0 degrees Fahrenheit [F] oral or equivalent) and/or clinically significant respiratory illness (example, cough or sore throat) within 14 days prior to randomization
* Any known immunosuppressive condition or immune deficiency disease, including human immunodeficiency virus infection, or ongoing immunosuppressive therapy
* History of Guillain-Barré syndrome

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 301 (Actual)
Dates: Start 2015-06; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ashwin Swami, MD, Study Director — MedImmune LLC
Locations (3):
- United States (3):
  - Research Site, South Miami, Florida
  - Research Site, Stockbridge, Georgia
  - Research Site, Portland, Oregon

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 300 participants were randomized and participated in the study from 15-Jun-2015 through 15-Jan-2016 at 3 sites in the United States of America (USA).
Groups:
- Placebo: Participants received a single dose of placebo matching with trivalent influenza vaccine by intranasal spray on Day 1.
- Trivalent Influenza Vaccine: Participants received a single dose of trivalent influenza vaccine [10^7.0 +/- 0.5 fluorescent focus unit (FFU) of each of 3 cold adapted (ca), attenuated (att), temperature sensitive (ts) 6:2 reassortant influenza strains] by intranasal spray on Day 1.
Period: Overall Study
Arm/Group | Placebo | Trivalent Influenza Vaccine
Started | 60 | 240
Completed | 59 | 238
Not Completed | 1 | 2
Not completed — Lost to Follow-up | 1 | 2

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) population included all participants that were randomized and treated with investigational product.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Trivalent Influenza Vaccine | Total
Number analyzed (Participants) | 60 | 240 | 300
Age, Continuous [Mean (Standard Deviation); unit: Years] | 30.2 (9.2) | 32.3 (9.5) | 31.9 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 136 | 164
  Male | 32 | 104 | 136

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Fever Greater Than or Equal to (>=) 101 Degrees Fahrenheit (F)
Description: Percentage of participants with fever defined as oral temperature >=101 degrees F were reported.
Time Frame: Baseline (Day 1) up to Day 8
Population: as for baseline characteristics
Measure: Number; unit: Percentage of Participant
Arm/Group | Placebo | Trivalent Influenza Vaccine
Number analyzed (Participants) | 60 | 240
Percentage of Participant | 0 | 0.4
Statistical Analysis 1: Comparison: Placebo vs Trivalent Influenza Vaccine; Test type: Superiority or Other; Rate Difference = 0.4, 95% CI 2-sided [-5.2 to 2.6]

2. Secondary Outcome: Percentage of Participants With Solicited Symptoms
Description: Solicited symptoms are predefined symptoms or events specifically inquired about and assessed daily after vaccine administration up to 15 days after vaccination. The solicited symptoms include fever greater than (>) 100.0 degrees F (37.8 degrees Celsius), runny nose, sore throat, cough, vomiting, muscle aches, chills, decreased activity and headache. Results were reported for all solicited symptoms except fever >=101 degrees F (reported as primary outcome) within 8 days after vaccination and all solicited symptoms within 15 days after vaccination.
Time Frame: Baseline (Day 1) up to Day 8 and Day 15
Population: The ITT population included all participants that were randomized and treated with investigational product.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Trivalent Influenza Vaccine
Number analyzed (Participants) | 60 | 240
Percentage of Participants
  Up to Day 8 | 20.0 | 36.7
  Up to Day 15 | 21.7 | 39.6
Statistical Analysis 1: Comparison: Placebo vs Trivalent Influenza Vaccine; Up to Day 8; Test type: Superiority or Other; Rate Difference = 16.7, 95% CI 2-sided [3.6 to 27.6]
Statistical Analysis 2: Comparison: Placebo vs Trivalent Influenza Vaccine; Up to Day 15; Test type: Superiority or Other; Rate Difference = 17.9, 95% CI 2-sided [4.4 to 29.3]

3. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Treatment-emergent AEs were events between administration of study drug and up to 15 days after vaccination that are absent before treatment or that worsened relative to pre-treatment state. Results were given for AEs reported within 8 days and 15 days after vaccination.
Time Frame: Baseline (Day 1) up to Day 8 and Day 15
Population: The ITT population included all participants that were randomized and treated with investigational product.
Measure: Number; unit: Participants
Arm/Group | Placebo | Trivalent Influenza Vaccine
Number analyzed (Participants) | 60 | 240
Participants
  Up to Day 8 | 3 | 13
  Up to Day 15 | 3 | 14

4. Secondary Outcome: Number of Participants With Treatment Emergent Serious Adverse Events (TESAEs) and New Onset Chronic Disease (NOCDs)
Description: An AE is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent SAEs were serious events between administration of study drug and up to 181 days after the dose that are absent before treatment or that worsen relative to pretreatment state. An NOCD is a newly diagnosed medical condition that is of a chronic, ongoing nature and is assessed by the investigator as medically significant. Results were given for TESAEs and NOCDs reported within 29 days and 181 days after vaccination.
Time Frame: Baseline (Day 1) up to Day 29 and 181
Population: The ITT population included all participants that were randomized and treated with investigational product.
Measure: Number; unit: Participants
Arm/Group | Placebo | Trivalent Influenza Vaccine
Number analyzed (Participants) | 60 | 240
Participants
  Up to Day 29: TESAEs | 0 | 0
  Up to Day 29: NOCDs | 0 | 0
  Up to Day 181: TESAEs | 0 | 1
  Up to Day 181: NOCDs | 0 | 0

5. Secondary Outcome: Percentage of Participants Who Require Antipyretic and/or Analgesic Medication
Description: Percentage of participants who require antipyretic and/or analgesic medication were reported.
Time Frame: Baseline (Day 1) up to Day 8 and Day 15
Population: The ITT population included all participants that were randomized and treated with investigational product.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Trivalent Influenza Vaccine
Number analyzed (Participants) | 60 | 240
Percentage of Participants
  Up to Day 8 | 0 | 0.4
  Up to Day 15 | 0 | 0.8

ADVERSE EVENTS:
Time Frame: Adverse Events: From Screening (Day -14) up to Day 15, and Serious Adverse Events: From Screening (Day -14) up to Day 181
Arm/Group | Placebo | Trivalent Influenza Vaccine
Serious Adverse Events (participants affected / at risk) | 0/60 | 1/240
Other Adverse Events (participants affected / at risk) | 3/60 | 14/240
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=60) | Trivalent Influenza Vaccine (N=240)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=60) | Trivalent Influenza Vaccine (N=240)
Lacrimation increased (Eye disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hordeolum (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 1 (1)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (5)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome. The PIs also agree for data to be presented first as a joint, multi-center publication.